CLINICAL TRIAL: NCT01498575
Title: An Evaluation of a Web-based Intervention Program for Parents and Teens to Promote Safe Driving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: State Farm Insurance Co. (Unknown); Bryn Mawr Rehabilitation Hospital (Unknown); GFK Knowledge Networks (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11-008203
Record Dates: First submitted 2011-12-20; First posted 2011-12-23 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Novice Teen Driver Training
Keywords: Teen driving; Behind the wheel practice driving; Parent supervision

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teen Driving Plan (Experimental): Access to web-based driving intervention
  Interventions: Behavioral: Teen driving plan
- Usual practice (No Intervention): Use of typical supervised practice driving resources

INTERVENTIONS:
Behavioral: Teen driving plan — Web-based intervention designed to facilitate parent supervised practice driving with novice teen driver.
  Arms: Teen Driving Plan

SUMMARY:
The long-term goal of this research is to increase safe driving among novice teen drivers by increasing the quantity, quality and diversity of driving practice while accompanied by an adult. In order to achieve the long term goal of the study, the investigators have developed a web-based intervention program known as Teen Driving Plan (TDP) intended to support high quality driving practice.

DETAILED DESCRIPTION:
Motor vehicle crashes remain the number one cause of death among teens in the United States. Teen drivers (ages 16 to 19) are four times more likely to be involved in fatal crashes than adult drivers (ages 25 to 69). Inexperience is a fundamental factor in the high crash rate for novice teens. Safe and skilled driving is a complex task that involves behaviors (e.g., skills and actions) that vary and become increasingly challenging with increasing speed, unsafe road conditions and other hazards of the driving environment. Because teens are at their lowest lifetime risk of crashing when accompanied by an adult, adult-supervised practice provides a safe way for teens to gain needed experience under a variety of driving conditions. Unfortunately, few teens receive sufficient quantity, quality and diversity of adult-supervised practice prior to licensure.

The objective of the proposed research is to compare how the driving training process and the results of that training process differ between a group of young learning permit holders in families that have access to TDP (the intervention group) from the training process and the results of that process in an otherwise similar group of teens in families with no TDP access (the control group). The investigators hypothesize that teens given access to TDP will demonstrate greater competence and safety in a standardized on-road driving assessment than teens with no TDP access.

ELIGIBILITY:
Inclusion Criteria:

* Teen 16 or 17 years of age who holds a Pennsylvania (PA) learner permit, or plans to obtain a learner permit in < 1 month.
* Parent(s) or legal guardian(s) of a teen with his or her learner permit.
* Internet connection at home and other technical requirements to launch web program if needed.

Exclusion Criteria:

* Non-English speaking.
* Teen has practiced more than 5 hours behind the wheel or has taken more than 5 practice drives with a supervising adult prior to enrollment.
* Teen has received formal behind-the-wheel driver education instruction prior to enrollment with a certified driving instructor at a professional driver education company or in his/her school.
* Pregnant female teen subjects.
* Teen requires handicapped placard or license plate in order to drive.

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1024 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis R Durbin, MD, MSCE, Principal Investigator — Chidlren's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Mirman JH, Curry AE, Winston FK, Wang W, Elliott MR, Schultheis MT, Fisher Thiel MC, Durbin DR. Effect of the teen driving plan on the driving performance of teenagers before licensure: a randomized clinical trial. JAMA Pediatr. 2014 Aug;168(8):764-71. doi: 10.1001/jamapediatrics.2014.252. PMID 24957844
- [Derived] Winston FK, Mirman JH, Curry AE, Pfeiffer MR, Elliott MR, Durbin DR. Engagement with the TeenDrivingPlan and diversity of teens' supervised practice driving: lessons for internet-based learner driver interventions. Inj Prev. 2015 Feb;21(1):4-9. doi: 10.1136/injuryprev-2014-041212. Epub 2014 Jun 10. PMID 24916684

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From December 2011 to August 2012, participants were recruited from 5 sources: (1) local high schools; (2) The Children's Hospital of Philadelphia (CHOP) primary care practices; (3) local licensing centers; (4) community events; and (5) targeted ads in online venues. Fliers, letters, and ads describing the study were distributed via these channels.
Pre-assignment Details: A subset of the teens were assigned to complete the On Road Driving (ODA) assessment. Study participation lasted from 6-36 months based on licensure status - all dyads participated in the study for 6 months, after which participation continued until teens obtained their junior driver's license (up to a max of 36 months from enrollment).
Groups:
- Teen Driving Plan (TDP): Access to web-based driving intervention
  Teen driving plan: Web-based intervention designed to facilitate parent supervised practice driving with novice teen driver.
- Usual Practice (Control): Use of typical supervised practice driving resources
Period: Overall Sample
Arm/Group | Teen Driving Plan (TDP) | Usual Practice (Control)
Started | 610 | 414
Completed | 550 | 400
Not Completed | 60 | 14
Not completed — Withdrawal by Subject | 60 | 14
Period: On the Road Driving Assessment (ODA)
Arm/Group | Teen Driving Plan (TDP) | Usual Practice (Control)
Started | 128 | 89
Completed | 86 | 65
Not Completed | 42 | 24
Not completed — Withdrawal by Subject | 19 | 6
Not completed — Protocol Violation | 23 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teen Driving Plan | Usual Practice | Total
Number analyzed (Participants) | 610 | 414 | 1024
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Teens (n=315, 210) | 16.2 [16.1 to 16.6] | 16.3 [16.1 to 16.7] | 16.2 [16 to 17]
  Parents (n=295, 204) | 48.4 [44.7 to 51.8] | 48.9 [45.8 to 51.9] | 48.5 [45 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 385 | 278 | 663
  Male | 225 | 136 | 361
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 9 | 23
  Not Hispanic or Latino | 591 | 402 | 993
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 11 | 17 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 68 | 46 | 114
  White | 516 | 342 | 858
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Late Driving Performance in On-road Assessment (ODA) Test
Description: The primary outcome was driving performance as measured by the teens completion of the standardized and validated ODA 24 weeks after enrollment. Certified professional driving evaluators blinded to randomization status terminated the ODA if they determined that the teen could not safely complete it. Criteria for termination included: (1) a driver action or inaction requiring evaluator intervention to prevent a collision; (2) a driving task requiring assistance from the evaluator to be performed safely; (3) violation of a traffic law; (4) evasive action needed by another vehicle or a pedestrian to avoid a collision; or (5) a subjective assessment by the evaluator that the teenager could not continue safely. We examined the teens ability to complete the ODA as measured by the number of terminations.
Time Frame: 24 weeks after enrollment
Population: 512 teen-parent dyads were eligible and agreed to participate. Of these, 217 teens were scheduled to complete the ODA (128 were randomized to Teen Driving Plan (TDP), 89 to Usual Practice). Participant attrition over the time of the study resulted in 151 teens (86 TDP and 65 control) completing the 24-week ODA.
Measure: Number; unit: Participants
Groups:
- Teen Driving Plan (TDP): Access to web-based driving intervention that provides practice supervisors with specific guidance for facilitating supervision of teens' practice drives across several environments and conditions (eg., highways, commercial districts) using brief instructional videos and resources.
- Usual Practice (Control): Participants received a hard copy of the Pennsylvania driver's manual, also available online and at licensing centers.
Arm/Group | Teen Driving Plan (TDP) | Usual Practice (Control)
Number analyzed (Participants) | 86 | 65
Participants | 5 | 10

ADVERSE EVENTS:
Time Frame: 24 weeks from time of enrollment
Arm/Group | Teen Driving Plan (TDP) | Usual Practice (Control)
Serious Adverse Events (participants affected / at risk) | 0/610 | 0/414
Other Adverse Events (participants affected / at risk) | 0/610 | 0/414

LIMITATIONS AND CAVEATS:
Moderate attrition (although no evidence of selective attrition); limited generalizability of results; and eight teenagers were not administered the highway module and were censored from analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No